CLINICAL TRIAL: NCT04190394
Title: Comparison of Two Exercise Training Modalities on Left Myocardial Regional Function After MI (Myocardial Infarction) Evaluated by 2D Strain Ultrasound - a Randomized Controlled Bicentric Study
Brief Title: Comparison of Two Exercise Training Modes on Left Myocardial Regional Function After Myocardial Infarction Evaluated by 2D Strain Ultrasound
Acronym: STRAICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NIMAO/2018-03/AD-01
Record Dates: First submitted 2019-12-02; First posted 2019-12-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Cardiomyopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator will not know which group of patients the results are from.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients following the CONT program (No Intervention): In the " CONT continuous training" group, the control group, the patient benefits from a retraining program according to the continuous mode (see details in section 3.4) for 8 weeks, with three 40-minute sessions per week.
- Patients following the IT program (Experimental): In the "IT intermittent training group", group, (the experimental group), the patient benefits from a retraining program according to the intermittent mode (see details in section 3.4) for 8 weeks, with three 45-minute sessions per week.
  Interventions: Other: Intermittent retraining program.

INTERVENTIONS:
Other: Intermittent retraining program. — Patient benefits from an intermittent retraining program for 8 weeks, with three 45-minute sessions per week.
  Arms: Patients following the IT program

SUMMARY:
Ischemic cardiomyopathy, defined by a deficiency in oxygenation of the myocardium due to a narrowing of the coronary arteries, is a major problem for public health. Medicinally-treated or re-vascularized cardiovascular rehabilitation following myocardial infarction has shown undeniable benefits in decreasing the overall mortality rate (13-26%), cardiovascular mortality (26-36%) and morbidity, by controlling cardiovascular risk factors and improving tolerance to effort and consequently improving the quality of life. Since the integration of physical exercise into the rehabilitation programs of patients suffering from coronary disease in the mid-90s, and throughout the following decade, the exercise training program has mainly relied on moderately intense continuous exercises (CONT) the aim of which is to improve the aerobic capacity. These efforts typically consist of performing a submaximal exercise with an intensity of 50 to 80% of the maximum capacity for effort (established according to studies depending on the maximum or reserve heart rate or even peak power, measured when performing a first test, then a progressive and maximum test), and a constant duration (about 20 to 60 minutes). In the 2000s, under the aegis of Scandinavian teams, the intermittent mode (IT) appeared, characterized by alternating high intensity efforts of a short duration with active recuperation phases (Rognmo et al., 2004). Superiority of the IT mode over the CONT mode is generally observed on aerobic capacity for effort, usually gauged via the maximal oxygen consumption peak measured during a graded and maximum effort test. An important methodological bias in the comparison of the two modalities, within meta-analyses or even in the same randomized controlled trial, is the absence of control/pairing on the overall volume of training. At the present time, and to the best of our knowledge, there have been no studies to compare the effects of CONT versus IT modes on the systolic or diastolic function of the myocardial region by 2D-strain following myocardial infarction. The aim of our study was to compare the outcomes of 2D strain scans upon inclusion and after 8 weeks of cardiovascular physiotherapy for 2 groups of patients benefiting from a CONT or IT program.

DETAILED DESCRIPTION:
This is a bi-centric randomised comparative superiority trial, blinded to the evaluator for 2 parallel groups (interventional intermittent training group "IT" vs a continuous training control group "CONT") with a 1:1 ratio.

Patients admitted for care at the cardiology departments of Nîmes University Hospital and the cardiology department of Avignon hospital for a first myocardial infarction dating back to less than 6 weeks will be pre-selected. The patients will receive both written and oral information about the study.

Patients are then referred to the Physical Medicine and Cardiac Rehabilitation departments at Nîmes University Hospital for the Nîmes site and the Lavarin Cardio Rehabilitation Center for the Avignon site for the inclusion visit at which the information about the study is given. Patients will be included in the study after signing a consent form.

The investigators then proceed with a maximal aerobic exercise test to evaluate cardiovascular endurance capacities and the suitability of the cardiovascular training program. Cardiac ultrasound is also performed, questionnaires about the quality of life are administered and biological doses are measured.

Then a stratified randomisation on the patient's age and sex will be performed to assign the subject either to the "IT intermittent training group" group, the experimental group, or to the "CONT continuous training" group, the control group which corresponds to the general care usually given.

Comparison of these two groups constitutes the methodological framework for this research. In the "IT intermittent training group (the experimental group), the patient benefits from a retraining program according to intermittent mode for 8 weeks, with three 45-minute sessions per week.

In the "CONT continuous training" group (the control group), the patient benefits from a retraining program according to the continuous mode for 8 weeks, with three 40-minute sessions per week.

At the end of the retraining program, at 8 weeks, an exercise test and a 2D Strain scan are performed, biological doses are taken and quality of life questionnaires are handed out.

Each patient will be followed 2 months after inclusion. The duration of inclusion period will be 18 months. The total duration of the test will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* patient must have given free informed consent and signed the consent form
* patient must be affiliated to or be covered by a health insurance scheme.
* patient must be an adult aged ≥ 18 to ≤ 75 years old.
* Patient must have had a first episode of myocardial infarction treated via medical treatment or by revascularization like a percutaneous transluminal angioplasty (only if the patient has had complete revascularization) at least 6 weeks previously.

Exclusion Criteria:

* The patient is participating in another intervention study or has taken part in another interventional study in the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is often under curatorship, tutorship or advisorship.
* It is impossible to give the patient clear information
* The patient refuses to sign the consent form
* The patient is pregnant, about to give birth or breastfeeding
* The patient has a contraindication for retraining
* The patient has a prosthetic heart valve
* The patient has severe valve disorder
* The patient requires cardiac stimulation
* The patient has an automatic implantable defibrillator
* The patient has sinus tachycardia, sinus bradycardia or sinus arrhythmia
* The patient has non-controlled high blood pressure
* The patient has a ventricular ejection fraction < 45%
* The patient has already participated in a cardiac rehabilitation program less than a year before
* The patient has a relapse of myocardial ischaemia during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Longitudinal systolic strain on Day 0. | Day 0
  All patients, whatever group they have been assigned to, will undergo a 2D Strain scan at the inclusion visit, before starting continuous (CONT) or intermittent (IT) cardiovascular rehabilitation.The overall longitudinal systolic strain (s-1) of the left ventricle will be measured (%) by echocardiography.
Longitudinal systolic strain at Week 8. | Week 8
  All patients whatever group they have been assigned to will undergo a 2D Strain scan after undergoing 8 weeks continuous (CONT) or intermittent (IT) of cardiovascular physiotherapy.The overall longitudinal strain (s-1) of the left ventricle will be measured (%) by echocardiography.

SECONDARY OUTCOMES:
Longitudinal diastolic strain on Day 0 | D0
  Longitudinal diastolic strain (s-1) will be measured by echocardiography before undergoing CONT or IT cardiovascular rehabilitation.
Longitudinal diastolic strain at Week 8 | Week 8
  Longitudinal diastolic strain (s-1) will be measured by echocardiography after 8 weeks of CONT or IT cardiovascular rehabilitation.
Circumferential strain on Day 0 | Day 0
  Circumferential strain (s-1) will be measured by echocardiography before beginning CONT or IT cardiovascular rehabilitation.
Circumferential strain at Week 8 | Week 8
  Circumferential strain (s-1) will be measured by echocardiography after undergoing CONT or IT cardiovascular rehabilitation.
Systolic radial strain on Day 0 | Day 0
  Systolic radial strain (%) will be measured by echocardiography before beginning CONT or IT cardiovascular rehabilitation.
Systolic radial strain at Week 8 | Week 8
  Systolic radial strain (%) will be measured by echocardiography after undergoing CONT or IT cardiovascular rehabilitation.
Diastolic radial strain on Day 0 | Day 0
  Diastolic radial strain (s-1) will be measured by echocardiography before beginning CONT or IT cardiovascular rehabilitation.
Diastolic radial strain at Week 8 | Week 8
  Diastolic radial strain (S-1) will be measured by echocardiography after undergoing CONT or IT cardiovascular rehabilitation.
Systolic circumferential strain on Day 0 | D0
  Systolic circumferential strain (s-1) will be measured before undergoing CONT or IT cardiovascular rehabilitation.
Systolic circumferential strain at Week 8 | Week 8
  Systolic circumferential radial strain (s-1) will be measured after undergoing 8 weeks of CONT or IT cardiovascular rehabilitation.
Diastolic circumferential strain on Day 0 | Day 0
  Diastolic circumferential strain (s-1) will be measured before undergoing CONT or IT cardiovascular rehabilitation.
Diastolic circumferential strain at Week 8 | Week 8
  Diastolic circumferential strain (s-1) will be measured after undergoing CONT or IT cardiovascular rehabilitation.
Apical rotation on Day 0 | Day 0
  Apical rotation (°) will be measured before undergoing CONT or IT cardiovascular rehabilitation.
Apical rotation at Week 8 | Week 8
  Apical rotation (°) will be measured after undergoing 8 weeks of CONT or IT cardiovascular rehabilitation.
Basal rotation on Day 0 | Day 0
  Basal rotation (°) will be measured before undergoing CONT or IT cardiovascular rehabilitation.
Basal rotation at Week 8 | Week 8
  Basal rotation (°) will be measured after undergoing 8 weeks of CONT or IT cardiovascular rehabilitation.
Ventricular torsion on Day 0 | Day 0
  Ventricular torsion (°) will be measured before undergoing CONT or IT cardiovascular rehabilitation.
Ventricular torsion at Week 8 | Week 8
  Ventricular torsion (°) will be measured after undergoing 8 weeks of CONT or IT cardiovascular rehabilitation.
Intraventricular asynchrony on Day 0 | Day 0
  Intraventricular asynchrony (ms) will be measured before undergoing CONT or IT cardiovascular rehabilitation.
Intraventricular asynchrony at Week 8 | Week 8
  Intraventricular asynchrony (ms) will be measured after undergoing 8 weeks of CONT or IT cardiovascular rehabilitation.
Cardiac morphology : Telesystolic volume on Day 0 | D0
  Telesystolic volume wil be measured (mL) before starting cardiac rehabilitation.
Cardiac morphology : Telesystolic volume at Week 8 | Week 8
  Telesystolic volume wil be measured (mL) after cardiac rehabilitation.
Cardiac morphology : Telediastolic volume on Day 0 | Day 0
  Telediastolic volume will be measured (mL) before starting cardiac rehabilitation.
Cardiac morphology : Telediastolic volume at Week 8 | Week 8
  Telediastolic volume will be measured (mL) after cardiac rehabilitation.
Cardiac morphology : Left ventricle mass on Day 0 | Day 0
  Left ventricle mass will be measured (g/m²) before starting cardiac rehabilitation.
Cardiac morphology : Left ventricle mass at Week 8 | Week 8
  Left ventricle mass will be measured (g/m²) after cardiac rehabilitation.
Cardiac morphology : FEVG at Day 0 | Day 0
  FEVG will be measured (%) before cardiac rehabilitation.
Cardiac morphology : FEVG at Week 8 | Week 8
  FEVG will be measured (%) after cardiac rehabilitation.
Cardiac morphology : S' wave on Day 0 | Day 0
  S' wave will be measured (%) before cardiac rehabilitation.
Cardiac morphology : S' wave at Week 8 | Week 8
  S' wave will be measured (%) after cardiac rehabilitation.
Cardiac morphology : E/A ratio on Day 0 | Day 0
  E/A ratio will be measured before cardiac rehabilitation.
Cardiac morphology : E/A ratio at Week 8 | Week 8
  E/A ratio will be measured after cardiac rehabilitation.
Cardiac morphology : E' wave at Day 0 | Day 0
  E' wave will be measured cm/s) before cardiac rehabilitation.
Cardiac morphology : E' wave at Week 8 | Week 8
  E' wave will be measured (cm/s) after cardiac rehabilitation.
Cardiac morphology : A' wave on Day 0 | Day 0
  A' wave will be measured (cm/s) before cardiac rehabilitation.
Cardiac morphology : A' wave at Week 8 | Week 8
  A' wave will be measured (cm/s) after cardiac rehabilitation.
Cardiac morphology : E/E' ratio on Day 0 | Day 0
  E/E' ratio will be measured before cardiac rehabilitation.
Cardiac morphology : E/E' ratio at Week 8 | Week 8
  E/E' ratio will be measured after cardiac rehabilitation.
Cardiac morphology : Systolic ejection volume on Day 0 | Day 0
  Systolic ejection volume will be measured before cardiac rehabilitation.
Cardiac morphology : Systolic ejection volume at Week 8 | Week 8
  Systolic ejection volume will be measured after cardiac rehabilitation.
Aerobic capacity: VO2max on Day 0 | Day 0
  VO2max (mL/min/kg) is measured with a Jaeger Oxycon Pro ergospirometer before starting cardiac rehabilitation.
Aerobic capacity: VO2max at Week 8 | Week 8
  VO2max (mL/min/kg) is measured with a Jaeger Oxycon Pro ergospirometer after undergoing 8 weeks of cardiac rehabilitation.
Aerobic capacity: Maximal aerobic power (MAP) on Day 0 | Day 0
  MAP (watts) is measured with a Jaeger Oxycon Pro ergospirometer before starting cardiac rehabilitation .
Aerobic capacity : Maximal aerobic power (MAP) at Week 8 | Week 8
  MAP (watts) is measured with a Jaeger Oxycon Pro ergospirometer after undergoing 8 weeks of cardiac rehabilitation .
Aerobic capacity: ventilation threshold (mL/min/kg) on Day 0 | Day 0
  The ventilation threshold VT1 (mL/min/kg) is measured with a Jaeger Oxycon Pro before starting cardiac rehabilitation.
Aerobic capacity: ventilation threshold (mL/min/kg) at Week 8 | Week 8
  The ventilation threshold VT1 (mL/min/kg) is measured with a Jaeger Oxycon Pro ergospirometer after undergoing 8 weeks of cardiac rehabilitation.
Aerobic capacity: walking on Day 0 | Day 0
  Performance at a 6-minute (m) walk is measured with a Jaeger Oxycon Pro ergospirometer before starting cardiac rehabilitation.
Aerobic capacity: walking at Week 8 | Week 8
  Performance at a 6-minute (m) walk is measured with a Jaeger Oxycon Pro ergospirometer after undergoing 8 weeks of cardiac rehabilitation.
Weight on Day 0 | Day 0
  The patient's weight will be measured in kilograms before beginning cardiac rehabilitation.
Weight at Week 8 | Week 8
  The patient's weight will be measured in kilograms after undergoing 8 weeks of cardiac rehabilitation.
Height on Day 0 | Day 0
  The patient's height will be measured in centimeters before beginning cardiac rehabilitation.
Height at Week 8 | Week 8
  The patient's height will be measured in centimeters after undergoing 8 weeks of cardiac rehabilitation.
Waist measurement on Day 0 | Day 0
  The patient's waist measurement will be noted in centimeters before beginning cardiac rehabilitation.
Waist measurement at Week 8 | Week 8
  The patient's waist measurement will be noted in centimeters after undergoing 8 weeks of cardiac rehabilitation.
Body Mass Index on Day 0 | Day 0
  The patient's Body Mass Index will be calculated in kg/m2 before beginning cardiac rehabilitation.
Body Mass Index at Week 8 | Week 8
  The patient's Body Mass Index will be calculated in in kg/m2 after undergoing 8 weeks of cardiac rehabilitation.
Medicinal treatment on Day 0 | Day 0
  Any medicinal treatment that the patient may be following will be noted before beginning cardiac rehabilitation.
Medicinal treatment at Week 8 | Week 8
  Any medicinal treatment that the patient may be following will be noted after undergoing 8 weeks of cardiac rehabilitation.
Hemoglobin in g/dL on Day 0 | Day 0
  A blood sample will be taken before beginning cardiac rehabilitation and Hemoglobin will be measured in g/dL.
Hemoglobin in g/dL at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Hemoglobin will be measured in g/dL.
Percentage volume of Hematocrit on Day 0 | Day 0
  A blood sample will be taken before beginning cardiac rehabilitation and Hematocrit will be measured as a percentage.
Percentage volume of Hematocrit at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Hematocrit will be measured as a percentage.
Mean Corpuscular Volume in femtoliters on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and Mean Corpuscular Volume will be measured in fL.
Mean Corpuscular Volume in femtoliters at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Mean Corpuscular Volume will be measured in fL.
Platelets in G/L on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and platelets will be measured in G/L.
Platelets in G/L at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and platelets will be measured in G/L.
Leukocytes in G/L on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and leukocytes will be measured in G/L.
Leukocytes in G/L at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and leukocytes will be measured in G/L.
C-reactive Protein on Day 0 | Day 0
  A blood sample will be taken before beginning cardiac rehabilitation and C-reactive Protein will be measured in mg/L.
C-reactive Protein at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and C-reactive Protein will be measured in mg/L.
Potassium in millimoles per liter on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and potassium will be measured in mmol/l.
Potassium in millimoles per liter at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and potassium will be measured in mmol/l.
Sodium in millimoles per liter on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and sodium will be measured in mmol/l.
Sodium in millimoles per liter at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and sodium will be measured in mmol/l.
Urea on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and urea will be measured in milligrams per deciliter.
Urea at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and urea will be measured in milligrams per deciliter.
Creatinine on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and creatinine will be measured in milligrams per deciliter.
Creatinine at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and creatinine will be measured in milligrams per deciliter.
Fasting glucose on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and fasting glucose will be measured in milligrams per deciliter.
Fasting glucose at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and creatinine will be measured in milligrams per deciliter.
HbA1c on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and HbA1c will be measured as a percentage.
HbA1c at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and HbA1c will be measured as a percentage.
Aspartate Aminotransferase on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and Aspartate Aminotransferase will be measured in units per liter.
Aspartate Aminotransferase at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Aspartate Aminotransferase will be measured in units per liter.
Alanine Aminotransferase on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and Alanine Aminotransferase will be measured in units per liter.
Alanine Aminotransferase at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Alanine Aminotransferase will be measured in units per liter.
Alkaline phosphatase on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and Alkaline phosphatase will be measured in units per liter.
Alkaline phosphatase at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Alkaline phosphatase will be measured in units per liter.
  , bilirubin,Gamma-glutamyltransferase, total cholesterol, Low Density Lipoprotein-cholesterol, High Density Lipoprotein-cholesterol, triglycerides, NT-proB-type Natriuretic Peptides, micro-RNA (miRNA-22, miRNA208-a and miRNA 423-5p).
Creatine phosphokinase on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation Creatine phosphokinase will be measured in units per liter.
Creatine phosphokinase at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Creatine phosphokinase will be measured in units per liter.
Bilirubin on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and bilirubin will be measured in milligrams per deciliter.
Bilirubin at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and bilirubin will be measured in milligrams per deciliter.
Gamma-glutamyltransferase on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and gamma-glutamyltransferase will be measured in units per liter.
Gamma-glutamyltransferase at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and Gamma-glutamyltransferase will be measured in units per liter.
Total cholesterol on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and total cholesterol will be measured in milligrams per deciliter.
Total cholesterol at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and bilirubin will be measured in milligrams per deciliter.
Low Density Lipoprotein-cholesterol on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and low density lipoprotein-cholesterol will be measured in milligrams per deciliter.
Low Density Lipoprotein-cholesterol at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and low density lipoprotein-cholesterol will be measured in milligrams per deciliter.
High Density Lipoprotein-cholesterol on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and high density lipoprotein-cholesterol will be measured in milligrams per deciliter.
High Density Lipoprotein-cholesterol at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and high density lipoprotein-cholesterol will be measured in milligrams per deciliter.
Triglycerides on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and triglycerides will be measured in milligrams per deciliter.
Triglycerides at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and triglycerides will be measured in milligrams per deciliter.
NT-proB-type Natriuretic Peptides on Day 0 | Day 0
  A blood sample will be taken before starting cardiac rehabilitation and NT-proB-type natriuretic peptides will be measured in picograms per milliliter.
NT-proB-type Natriuretic Peptides at Week 8 | Week 8
  A blood sample will be taken after undergoing cardiac rehabilitation for 8 weeks and NT-proB-type natriuretic peptides will be measured in picograms per milliliter.
Micro-RNA dosage (miRNA22, miRNA122, miRNA150, miRNA208 a/b and miRNA 423-5p) on Day 0 | Day 0
  Micro-RNAs (including, notably, miRNA22, miRNA122, miRNA150, miRNA208 a/b and miRNA 423-5p) dosed via reverse-transcriptase quantitative polymerase chain reaction (PCR). PCR consists of an organic extraction stage followed by immobilization of RNA on an apparatus to purify it before elution. PCR provides numerous copies of a chosen DNA sequence. Real time quantitative PCR provides the quantity of DNA at each amplification cycle thanks to SYBR® Green, an intercalating fluorescent DNA agent, which emits a quantity of fluorescence for each amplicon produced. Fluorescence is thus directly proportional to the quantity of DNA in the sample. RNA extractions will be made from 200 μL of plasma collected before the patient starts cardiac rehabilitation and analyzed by researchers at Aix-Marseille University - INSERM, UMR 1260 C2VN Center for Cardiovascular and Nutrition research. Frozen samples will be shipped from Nîmes and Avignon to Marseille by Cryoglobe package.
Micro-RNA dosage (miRNA22, miRNA122, miRNA150, miRNA208 a/b and miRNA 423-5p) at Week 8 | Week 8
  Micro-RNAs (including, notably, miRNA22, miRNA122, miRNA150, miRNA208 a/b and miRNA 423-5p) dosed via reverse-transcriptase quantitative polymerase chain reaction (PCR). PCR consists of an organic extraction stage followed by immobilization of RNA on an apparatus to purify it before elution. PCR provides numerous copies of a chosen DNA sequence. Real time quantitative PCR provides the quantity of DNA at each amplification cycle thanks to SYBR® Green, an intercalating fluorescent DNA agent, which emits a quantity of fluorescence for each amplicon produced. Fluorescence is thus directly proportional to the quantity of DNA in the sample. RNA extractions will be made from 200 μL of plasma collected after the patient has had 8 weeks of cardiac rehabilitation and analyzed by researchers at Aix-Marseille University - INSERM, UMR 1260 C2VN Center for Cardiovascular and Nutrition research. Frozen samples will be shipped from Nîmes and Avignon to Marseille by Cryoglobe package.
Quality of life according to the WHOQOL-BREF Questionnaire on Day 0 | Day 0
  Before starting cardiac rehabilitation, the patient's quality of life is measured with the WHOQOL-BREF, a short version of the WHOQOL-100 quality of life assessment developed by the WHOQOL group with fifteen international field centres, simultaneously (Orley & Kuyken, 1994; Szabo, 1996; WHOQOL Group 1994a, 1994b, 1995). The WHOQOL-BREF questionnaire contains two items from the Overall QOL and General Health and 24 items of satisfaction divided into four domains: Physical health with 7 items (DOM1), psychological health with 6 items (DOM2), social relationships with 3 items (DOM3) and environmental health with 8 items (DOM4). Each item is rated on a 5-point Likert scale.The four domain scores denote an individual's perception of quality of life in each particular domain. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score.
Quality of life according to the WHOQOL-BREF Questionnaire at Week 8 | Week 8
  After undergoing cardiac rehabilitation for 8 weeks, the patient's quality of life is measured with the WHOQOL-BREF, a short version of the WHOQOL-100 quality of life assessment developed by the WHOQOL group with fifteen international field centres, simultaneously (Orley & Kuyken, 1994; Szabo, 1996; WHOQOL Group 1994a, 1994b, 1995). The WHOQOL-BREF questionnaire contains two items from the Overall QOL and General Health and 24 items of satisfaction divided into four domains: Physical health with 7 items (DOM1), psychological health with 6 items (DOM2), social relationships with 3 items (DOM3) and environmental health with 8 items (DOM4). Each item is rated on a 5-point Likert scale.The four domain scores denote an individual's perception of quality of life in each particular domain. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score.
Quality of life according to the MacNew Questionnaire at Day 0 | Day 0
  Before starting cardiac rehabilitation, the patient's quality of life is measured with the MacNew Questionnaire, which is a self-administered modified version of the original QLMI instrument. The MacNew is designed to assess the patient's feelings about how Myocardial Infarction affects daily functioning and contains 27 items with a global Health-Related Quality of Life (HRQoL) score and subscales regarding physical limitation, emotional, and social function. There are 5 items that inquire about symptoms: angina/chest pain, shortness of breath, fatigue, dizziness, and aching legs.The items and scales are scored from 1 (low HRQoL) to 7 (high HRQoL), and the minimal important difference on each MacNew scale is 0.50 points. The time frame for the MacNew is the previous two weeks.
Quality of life according to the MacNew Questionnaire at Week 8 | Week 8
  After undergoing cardiac rehabilitation for 8 weeks, the patient's quality of life is measured with the MacNew Questionnaire, which is a self-administered modified version of the original QLMI instrument.The MacNew is designed to assess the patient's feelings about how Myocardial Infarction affects daily functioning and contains 27 items with a global Health-Related Quality of Life (HRQoL) score and subscales regarding physical limitation, emotional, and social function. There are 5 items that inquire about symptoms: angina/chest pain, shortness of breath, fatigue, dizziness, and aching legs. The items and scales are scored from 1 (low HRQoL) to 7 (high HRQoL), and the minimal important difference on each MacNew scale is 0.50 points. The time frame for the MacNew is the previous two weeks.
Observance of the rehabilitation program | Day 0 to Week 8
  An attendance sheet must be filled in by all patients, each time they attend their rehabilitation session whether they are assigned to the the control group (CONT) with three 40-minute sessions per week or the experimental group doing intermittent training (IT) with three 45-minute sessions per week.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud DUPEYRON, Dr., Principal Investigator — CHU de Nîmes (Nîmes University Hospital)
Locations (2):
- France (2):
  - Nîmes University Hospital, Nîmes, Gard
  - Clinique Lavarin, Centre de Rééducation Cardiaque,1 Rue Mère Térésa,, Avignon, Vaucluse

REFERENCES:
- [Result] Obert P, Nottin S, Belvisi C, Robert C, Miramont V, de France C, Carlioz R, Landrier JF, Poirier P, Dupeyron A. A comprehensive analysis of the impact of high-intensity interval vs. moderate-intensity continuous training on global and regional myocardial function in patients early after acute myocardial infarction - the STRAICT randomized controlled trial. Eur J Prev Cardiol. 2025 Mar 5:zwaf127. doi: 10.1093/eurjpc/zwaf127. Online ahead of print. PMID 40042823